CLINICAL TRIAL: NCT04134169
Title: A Multi-center, Open, Long-term Follow-up Study to Evaluate the Efficacy and Safety of FURESTEM-RA Inj. in Patients With Moderate to Severe Rheumatoid Arthritis : 5-year Results From the K0202 Extension Study
Brief Title: Long-term Observational Study to Evaluation the Safety of FURESTEM-RA Inj(K0202)
Status: Recruiting | Type: Observational
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: K0202-E
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis
  Interventions: Other: Not applicable(observational study)

INTERVENTIONS:
Other: Not applicable(observational study) — Not applicable(observational study)

SUMMARY:
Long-term Observational Study to Evaluation the Safety of FURESTEM-RA Inj(K0202)

DETAILED DESCRIPTION:
A Multi-center, Open, Long-term Follow-up Study to Evaluate the Efficacy and Safety of FURESTEM-RA Inj. in Patients With Moderate to Severe Rheumatoid arthritis: 5-year Results From the K0202 Extension Study

ELIGIBILITY:
Inclusion Criteria:

1. Subject who enrolled K0202 Clinical Trial(parent study) and has been given more than one medication.
2. Subjects who understand and voluntarily sign an informed consent form

Exclusion Criteria:

1. Any other condition which the investigator judges would make patient unsuitable for study participation

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to Severe Rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2025-08-11 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment | 5 years
  (Rate of Adverse Event, Number of Participants with Adverse Event)

SECONDARY OUTCOMES:
1. Efficacy as measured by ACR(American College of Rheumatology)20,50,70 reaction rate | 5 years
2. Efficacy as measured by EULAR (European League Against Rheumatism)reaction rate | 5 years
change in DAS(Disease activity scores)28-ESR from baseline | 5 years
  DAS range is from ≥ 3.2 (inactive) , >3.2 but ≤ 5.1(moderate), >5.1(very active)
change in KHAQ(Korean Health assessment questionnaire) from baseline | 5 years
  KHAQ range is from 0 (clear) to 60 (severe)
change in CDAI (clinical disease activity index) from baseline | 5 years
  CDAI range is from 0 (clear) to 76 (severe)
change in 100mm Pain VAS(Visual analogue scale) from baseline | 5 years
  100mm Pain VAS range is from 0 (clear) to 100 (severe)
change in Modified Sharp/Van der Heijde Socre from baseline | 5 years
  Modified Sharp/Van der Heijde Socre range is from 0 (clear) to 448 (severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national University Boramae medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided